CLINICAL TRIAL: NCT05166681
Title: Evaluation of Surgical Wound Closure With Single Subcutaneous and Subdermal Sutures as a Single Layer in Comparison With Traditional Multiple Layer Closure in Plastic Surgery Procedures: A Randomized Controlled Trial
Brief Title: Evaluation of Aesthetic Surgical Wound Closure by a Single Layer in Comparison With Traditional Multi-layer Closure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abouqir General Hospital (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abouzaid, Dr. Ahmed Mohamed Abouzaid, Abouqir General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0304744
Record Dates: First submitted 2021-12-09; First posted 2021-12-22 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Surgical Wound Closure Technique
Keywords: surgical wound closure; subdermal wound suturing; traditional wound closure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): cases allocated to that arm are those cases having their surgical wound closure by the traditional techniques involving subcutaneous layer closure as one or more raws of sutures and then skin layer closure
  Interventions: Procedure: surgical wound suturing
- Single layer wound closure group (Experimental): cases allocated to that group are those having their surgical wound closure with the new technique involving part of the subcutaneous layer and the subdermal layer
  Interventions: Procedure: surgical wound suturing

INTERVENTIONS:
Procedure: surgical wound suturing — single layer surgical wound suturing in comparison with the traditional multi-layer wound suturing
  Other Names: single layer wound closure

SUMMARY:
the study is comparing the results of aesthetic surgery wound closure by a single layer versus the traditional multi-layer closure as regards the wound healing time, local wound complications, and the scar formed.

DETAILED DESCRIPTION:
The study puts in comparison the surgical wound closure of aesthetic procedures by single layer sutures technique, involving part of the subcutaneous tissue and the subdermal layer, with the multi-layer traditional closure, which involves subcutaneous layer closure by one or two raws of sutures and skin closure with any type of suturing techniques, then to evaluate the wound healing time, local wound complications, and the scar formed.

ELIGIBILITY:
Inclusion Criteria:

* all cases presented for different aesthetic surgery procedures e.g different breast contouring procedures, surgical trunk contouring procedures, Brachioplasty, and thigh lifting. No gender discrimination, age between 16-60 years.

Exclusion Criteria:

* we excluded cases in age groups beyond that designed for the study, patients with co-morbid conditions that may affect the results of wound healing e.g Diabetics. Active smokers, trauma patients, or patients that will undergo primary or secondary reconstructive procedures.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
single layer closure is as efficient and reliable as the multi-layer closure | 6 months follow up post-surgical
  single layer surgical wound closure is a reliable and efficient method as the traditional multi-layer closure technique giving the same results and have the same complication rate as the traditional suturing techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Abouqir General Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
data collected and results of the study will be evaluated and announced